CLINICAL TRIAL: NCT02232425
Title: An 8-Week, Double-Blind, Placebo-Controlled Parallel Group Study to Evaluate the Effect of IX-01 on Intravaginal Ejaculatory Latency Time (IELT) and Patient Reported Outcomes in Men With Lifelong Premature Ejaculation
Brief Title: IX-01 Effect on Intravaginal Ejaculatory Latency Time (IELT) and Patient Reported Outcomes in Men With Premature Ejaculation (PE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ixchelsis Limited (Industry)
Collaborators: Carelon Research (Other); Novotech (Australia) Pty Limited (Industry); ICON plc (Industry); PHT Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IX-0103
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Results first posted 2019-01-24 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: IX-01 (Experimental): Two to four 200 mg capsules administered orally, 1-6 hours prior to sexual activity
  Interventions: Drug: IX-01
- Placebo (Placebo Comparator): Two to four capsules administered orally, 1-6 hours prior to sexual activity
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IX-01
  Arms: Drug: IX-01
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effectiveness of IX-01 in men with lifelong premature ejaculation.

ELIGIBILITY:
Inclusion Criteria:

* In stable (≥ 6 months) heterosexual relationship
* Have life-long (primary) premature ejaculation
* Have premature ejaculation confirmed by Intravaginal Ejaculatory Latency Time (IELT) less than or equal to (≤) 1 minute on ≥ 75% attempts at sexual intercourse
* Meet other aspects of the International Society for Sexual Medicine (ISSM) definition for lifelong premature ejaculation (PE), including inability to delay ejaculation on all or nearly all vaginal penetrations and negative personal consequences such as distress, bother and frustration
* Willing to attempt intercourse at least 4 times during run-in period and at least 8 more times during double-blind part of the study
* Not planning pregnancy with his partner and he is willing to use contraception (unless not of child-bearing potential, e.g., surgically sterilised)
* Willing to limit use of alcohol on days in which they take study drug (not more than three drinks, where one drink is defined as a 12 ounce (oz), 360 milliliter (mL) bottle of beer, a 5 oz (150 mL) glass of wine, or a 1½ oz (45 mL distilled spirits)
* Capable of giving written informed consent

Exclusion Criteria:

* An Intravaginal Ejaculatory Latency Time (IELT) value ≥ 2 minutes during run-in period
* Less than (<) 4 attempts at sexual intercourse during run-in (screening may be extended or patient may be rescreened if there are extenuating circumstances)
* A rating of control of ejaculation as fair, good, or very good on the Premature Ejaculation Profile (PEP) questionnaire prior to study
* Co-existing Erectile Dysfunction - International Index of Erectile Dysfunction (IIEF) erectile function domain < 22 during run-in
* Concomitant use of Phosphodiesterase 5 (PDE5) inhibitors, intracavernosal injections, penile implants, Selective Serotonin Reuptake Inhibitors (SSRI's) or Serotonin-Norepinephrine Reuptake Inhibitors (SSNRI's), tricyclic antidepressants (for example (e.g.) clomipramine), monoamine oxidase inhibitors, alpha blockers, 5 alpha reductase inhibitors (including propecia for hair loss), topical anaesthetics, and/or tramadol
* History (last 6 months) of use of Botox or similar product to treat premature ejaculation
* Unwilling to stop other treatments for premature ejaculation (including but not limited to pharmacological, herbal, multiple condoms, psychosexual treatment, prior masturbation)
* Other sexual disorder of patient or partner that could interfere with results
* Current active sexually transmitted disease
* Major medical condition of patient that could interfere with ability to have sexual activity and or require hospital treatment
* Body Mass Index (BMI) > 40 kg/m2
* Participation in a clinical drug trial anytime during the 30 days prior to screening
* Human Immunodeficiency Virus (HIV) or hepatitis B
* History of clinically significant prostate disease
* History of myocardial infarction, coronary bypass surgery, coronary artery angioplasty, unstable angina, clinically evident congestive heart failure, cardiac pacemaker, or cerebrovascular accident
* Cardiac arrhythmia: significant cardiac arrhythmia shown on Electrocardiogram (ECG), or a known or suspected history of significant cardiac arrhythmias within last six months
* History of congenital QT prolongation and/ corrected QT (QTc) interval > 450 milliseconds (msec) using the Bazett formula
* Mean systolic cuff blood pressure (BP) > 140 millimeter of mercury (mmHg), as assessed by up to three measurements taken in sequence within 5-10 minutes of last measure
* Mean diastolic cuff BP > 90 mmHg, as assessed by up to three measurements taken in sequence within 5-10 minutes of the last measure
* Major psychiatric disease or risk of suicidal tendency as assessed by clinical evaluation and Patient Health Questionnaire (PHQ)-9 and Columbia Suicide Assessment
* PHQ-9 questionnaire total score > 9 and/or score > 0 for question 9 of PHQ-9, and/or suicidal ideation or behavior as assessed by Columbia Suicide Assessment
* Clinically significant abnormal laboratory function test results (including liver enzymes > 2 x Upper Limit of Normal (ULN) or bilirubin > 1.5 x ULN)
* Taking Cytochrome P450 3A4 (CYP3A4) inducers, or moderate and potent CYP3A4 inhibitors

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email Katie.George@Ixchelsis.com, Study Director — Ixchelsis Limited
Locations (10):
- United States (8):
  - San Diego Sexual Medicine, San Diego, California
  - South Florida Medical Research Inc., Aventura, Florida
  - Center for Marital and Sexual Health of South Florida, West Palm Beach, Florida
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Cooper Research Institute, Camden, New Jersey
  - Manhattan Medical Research, New York, New York
  - Urologic Consultants of Southeastern Pennsylvania, Bala-Cynwyd, Pennsylvania
  - Miriam Hospital / The Men's Health Center, Providence, Rhode Island
- Australia (2):
  - Australian Centre for Sexual Health, Saint Leonards, New South Wales
  - Keogh Institute for Medical Research, Nedlands, Western Australia

REFERENCES:
- [Derived] McMahon C, Althof S, Rosen R, Giuliano F, Miner M, Osterloh IH, Muirhead GJ, Harty B; PEPIX Multi-Centre Study Group. The Oxytocin Antagonist Cligosiban Prolongs Intravaginal Ejaculatory Latency and Improves Patient-Reported Outcomes in Men with Lifelong Premature Ejaculation: Results of a Randomized, Double-Blind, Placebo-Controlled Proof-of-Concept Trial (PEPIX). J Sex Med. 2019 Aug;16(8):1178-1187. doi: 10.1016/j.jsxm.2019.05.016. PMID 31351659

RESULTS

PARTICIPANT FLOW:
Groups:
- Drug: IX-01: Two to four 200 mg capsules administered orally, 1-6 hours prior to sexual activity
  IX-01
- Placebo: Two to four capsules administered orally, 1-6 hours prior to sexual activity
  Placebo
Period: Overall Study
Arm/Group | Drug: IX-01 | Placebo
Started | 58 | 30
Completed | 44 | 22
Not Completed | 14 | 8
Not completed — Lost to Follow-up | 6 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 5 | 6
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug: IX-01 | Placebo | Total
Number analyzed (Participants) | 58 | 30 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (9) | 43 (8) | 43 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 58 | 30 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 2 | 12
  Not Hispanic or Latino | 48 | 28 | 76
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 48 | 21 | 69
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 47 | 23 | 70
  Australia | 11 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean Fold Change in Geometric Mean Intravaginal Ejaculatory Latency Time (IELT)
Description: IX-01 versus placebo. Intravaginal ejaculatory latency time (IELT) was defined as the time from the initiation of sexual intercourse (penetration) until ejaculation occurred
Time Frame: Last 4 weeks of treatment compared to baseline
Population: Efficacy data set excluding outliers
Measure: Geometric Mean (95% Confidence Interval); unit: No units for fold change
Arm/Group | Drug: IX-01 | Placebo
Number analyzed (Participants) | 54 | 25
No units for fold change | 2.1 [1.5 to 3.1] | 1.1 [0.7 to 1.8]

2. Secondary Outcome: Proportion of Participants Rating Their PE as Better or Much Better, on the Clinical Global Impression of Change (CGIC) Scale
Description: 7 point scale ranging from much worse (-3) to much better (3). The proportion refers to the proportion of patients who had the best 2 possible responses [better(2) or much better (3)] on this 7 point scale
Time Frame: Baseline to the end of treatment (approximately 8 weeks)
Population: Intent to treat, excluding outliers
Measure: Number; unit: proportion of participants
Arm/Group | Drug: IX-01 | Placebo
Number analyzed (Participants) | 48 | 24
proportion of participants
  Better/Much Better | 0.17 | 0
  Any Improvement | 0.44 | 0.13

3. Secondary Outcome: Proportion of Participants With Greater Than or Equal to (≥) 2.5 Fold Increase in Intravaginal Ejaculatory Latency Time (IELT)
Description: Intravaginal ejaculatory latency time (IELT) was defined as the time from the initiation of sexual intercourse (penetration) until ejaculation occurred. Outcome measured proportion of patients with at least a 2.5-fold increase in geometric mean IELT over the last 4 weeks of treatment as compared to baseline. Proportion of participants adjusted for baseline IELT, country and site
Time Frame: Last 4 weeks of treatment compared to baseline
Population: Intent to treat, excluding outliers
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Drug: IX-01 | Placebo
Number analyzed (Participants) | 55 | 29
Proportion of participants | 0.31 [0.14 to 0.54] | 0.07 [0.01 to 0.32]

4. Secondary Outcome: Mean Fold Change in Arithmetic IELT (Intravaginal Ejaculatory Latency Time)
Description: IX-01 versus placebo
Time Frame: Last 4 weeks of treatment compared to baseline
Population: Intent to treat, excluding outliers
Measure: Mean (95% Confidence Interval); unit: No units for fold change
Arm/Group | Drug: IX-01 | Placebo
Number analyzed (Participants) | 54 | 25
No units for fold change | 3.6 [2.2 to 5.0] | 1.8 [0.9 to 2.7]

5. Secondary Outcome: Mean Change in Score on Control of Timing of Ejaculation
Description: Reported in electronic diary and based on the Premature Ejaculation Profile (PEP). PEP question on control of timing is scored on a 5 point scale with the scores ranging from very poor (this is the worst answer) scored as 0 to very good (this is the best answer scored as 4)
Time Frame: Last 4 weeks of treatment compared to baseline
Population: Intent to treat, excluding outliers
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Drug: IX-01 | Placebo
Number analyzed (Participants) | 54 | 25
units on a scale | 0.42 [-0.08 to 0.93] | -0.03 [-0.59 to 0.53]

6. Secondary Outcome: Mean Change in Score on Ejaculation-related Personal Distress
Description: Based on Premature Ejaculation Profile (PEP). Scale ranges from 'extremely' (0) to 'not at all' (4). An increase in score from baseline indicates improvement.
Time Frame: Last 4 weeks of treatment compared to baseline
Population: Intent to treat, excluding outliers
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Drug: IX-01 | Placebo
Number analyzed (Participants) | 54 | 25
units on a scale | 0.63 [0.37 to 0.88] | 0.03 [-0.34 to 0.40]

7. Secondary Outcome: Proportion of Participants With ≥ 1 Category of Improvement in Satisfaction With Sexual Intercourse, on the Premature Ejaculation Profile (PEP) Questionnaire
Description: Based on Premature Ejaculation Profile (PEP) 5 point scale with the scores ranging from 0 (worse answer) to 4 (best answer).
Time Frame: Baseline to 8 weeks
Population: Intent to treat, excluding outliers
Measure: Number (95% Confidence Interval); unit: adjusted proportion of participants
Arm/Group | Drug: IX-01 | Placebo
Number analyzed (Participants) | 52 | 25
adjusted proportion of participants | 0.53 [0.33 to 0.72] | 0.30 [0.13 to 0.56]

8. Secondary Outcome: Proportion of Participants With ≥ 1 Category of Improvement in Control Over Ejaculation During Sexual Intercourse on the Premature Ejaculation Profile (PEP) Questionnaire
Description: Reported in electronic diary and based on the Premature Ejaculation Profile (PEP). PEP is scored on a 5 point scale with the scores ranging from 0 (worst answer) to 4 (best answer)
Time Frame: Baseline to 8 weeks
Population: Intent to treat, excluding outliers
Measure: Number (95% Confidence Interval); unit: adjusted proportion of participants
Arm/Group | Drug: IX-01 | Placebo
Number analyzed (Participants) | 52 | 25
adjusted proportion of participants | 0.56 [0.42 to 0.69] | 0.36 [0.19 to 0.58]

9. Secondary Outcome: Proportion of Participants With ≥ 1 Category of Improvement in Ejaculation-related Distress on the Premature Ejaculation Profile ( PEP) Questionnaire
Description: Reported in e-diary. Based on Premature Ejaculation Profile (PEP). Scale ranges from 'extremely' (0) to 'not at all' (4). An increase in score from baseline indicates improvement.
Time Frame: Baseline to 8 weeks
Population: Intent to treat, excluding outliers
Measure: Number (95% Confidence Interval); unit: adjusted proportion of participants
Arm/Group | Drug: IX-01 | Placebo
Number analyzed (Participants) | 52 | 25
adjusted proportion of participants | 0.60 [0.46 to 0.73] | 0.36 [0.19 to 0.57]

10. Secondary Outcome: Proportion of Participants With ≥ 1 Category of Improvement in Ejaculation-related Interpersonal Difficulty on the Premature Ejaculation Profile (PEP) Questionnaire
Description: as for outcome 9
Time Frame: Baseline to 8 weeks
Population: Intent to treat, excluding outliers
Measure: Number (95% Confidence Interval); unit: adjusted proportion of participants
Arm/Group | Drug: IX-01 | Placebo
Number analyzed (Participants) | 52 | 25
adjusted proportion of participants | 0.60 [0.45 to 0.72] | 0.48 [0.29 to 0.68]

11. Secondary Outcome: Proportion of Participants With ≥ 2 Category Increase in Control and ≥ 1 Category Decrease in Personal Distress on a Patient Reported Outcome (PRO) Measure
Description: Reported in e-diary. Based on Premature Ejaculation Profile (PEP). Each of the PEP questions is scored on a 5 point scale with the scores ranging from 0 (worst answer) to 4 (best answer)
Time Frame: Baseline to 8 weeks
Population: Intent to treat, excluding outliers
Measure: Number; unit: proportion of participants
Arm/Group | Drug: IX-01 | Placebo
Number analyzed (Participants) | 52 | 25
proportion of participants | 0.17 | 0

12. Secondary Outcome: Change in Percentage of Intercourse Attempts Lasting Longer Than 1 Minute From Baseline to Last 4 Weeks on Treatment
Description: 'Baseline' time period defined as Day -28 - Day 0. 'Last 4 Weeks' time period defined as the 28 days prior to last time subject took study drug and after Day 14.
  Analysis excludes two subjects from ITT population: #010-012 (placebo) and #888-018 (active). Adjusted for treatment, baseline IELT, baseline percentage, country and site.
Time Frame: Baseline to last 4 weeks on treatment
Population: Intent to treat, excluding outliers
Measure: Mean (95% Confidence Interval); unit: percentage of attempts
Arm/Group | Drug: IX-01 | Placebo
Number analyzed (Participants) | 54 | 25
percentage of attempts | 37.6 [17.8 to 57.3] | 13.5 [-9.1 to 36.2]

13. Secondary Outcome: Incidence of Treatment-emergent Adverse Events
Description: Number of participants with at least one treatment-emergent adverse event
Time Frame: Start of Treatment to end of study (approximately 10 weeks)
Population: Intent to treat, excluding outliers
Measure: Number; unit: participants
Arm/Group | Drug: IX-01 | Placebo
Number analyzed (Participants) | 56 | 30
participants | 12 | 9

ADVERSE EVENTS:
Description: Two patients did not take any study medication hence 56 reported and not 58
Arm/Group | Drug: IX-01 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/30
Other Adverse Events (participants affected / at risk) | 12/56 | 9/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Drug: IX-01 (N=56) | Placebo (N=30)
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Dry Mouth (Gastrointestinal disorders) | 1 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Peridontal inflammation (Gastrointestinal disorders) | 1 | 0
Feeling jittery (General disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 1
Lacerations (Injury, poisoning and procedural complications) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Laboratory test abnormal (Investigations) | 1 | 0
Metabolic function test abnormal (Investigations) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Libido decreased (Psychiatric disorders) | 1 | 0
Renal Colic (Renal and urinary disorders) | 0 | 1
Rhinitis, allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor may choose to collaborate on authorship, and sponsor's agent has 60-day review